CLINICAL TRIAL: NCT01794533
Title: Analgesic Efficacy of a Combination of Fentanyl and Lidocaine for Maxillary Infiltration in Teeth With Irreversible Pulpitis
Brief Title: Effect of Fentanyl on the Rate of Anesthesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, fatemeh khodaei, Resident of Endodontics, Islamic Azad University, Sanandaj
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18050
Record Dates: First submitted 2013-01-30; First posted 2013-02-20 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Painful Irreversible Pulpitis
Keywords: Irreversible Pulpitis; Infiltration injection; Fentanyl; Lidocaine
MeSH Terms: interventions — Lidocaine; Epinephrine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine with Epinephrine+ Normal saline (Placebo Comparator)
  Interventions: Drug: Lidocaine with Epinephrine+ Normal saline; Drug: Lidocaine with Epinephrine + fentanyl
- Lidocaine with Epinephrine + fentanyl (Active Comparator)
  Interventions: Drug: Lidocaine with Epinephrine+ Normal saline; Drug: Lidocaine with Epinephrine + fentanyl

INTERVENTIONS:
Drug: Lidocaine with Epinephrine+ Normal saline — local infiltration of 1.8 mL of 2% lidocaine containing 1:200,000 epinephrine along with 0.8 mL of 0.9% sterile normal saline solution
Drug: Lidocaine with Epinephrine + fentanyl — local infiltration of 1.8 mL of 2% lidocaine, containing 1:200,000 epinephrine along with 0.8 mL of fentanyl(40 µg)
  Other Names: Sublimaze,fentanil

SUMMARY:
Achievement of a deep and long-durated anesthesia is vital before most endodontic procedures; therefore, the investigators conducted this study to compare the local infiltration effect of epinephrine-containing lidocaine with/ without fentanyl on depth and duration of anesthesia in maxillary molars with painful irreversible pulpitis.

DETAILED DESCRIPTION:
This study was planned with a randomized double-blind, parallel design clinical trial on 64 healthy patients after taking into account some inclusion and exclusion criteria. The control group were received the mixture of normal saline and 2% lidocaine with 1:200,000 epinephrine and the experimental group were received the mixture of fentanyl and 2% lidocaine with 1:200,000 epinephrine. The depth and duration of pulpal anesthesia were evaluated with an electric pulp testing in 5-minute intervals during a period of 60 minutes and the pain intensity recorded in five times, before injection, after injection, during access cavity preparation, pulpotomy and pulpectomy using visual analog scale(VAS). All data were analyzed and compared using chi-squared and Mann-Whitney tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients were aged between 18 and 65 years with no systemic diseases categorized in the Class I ASA;
* Individuals requiring urgent root canal treatment of maxillary first or second molars;
* Hot painful teeth with irreversible pulpitis (moderate to severe spontaneous pain), with a positive response to thermal vitality tests (a long painful response to a cold test) and no clinical or radiographic signs or symptoms of acute or chronic apical periodontitis; and
* No history of taking analgesics in the previous 12 h.

Exclusion Criteria:

* Systemic conditions;
* Allergic reactions to opioids, benzodiazepines, barbiturates;
* Pregnancy and lactation; Contraindication of the use of epinephrine (such as unstable angina);
* Nonvital pulp after access cavity preparation

Ages: 18 Years to 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in depth of anesthesia | Change from Baseline up to 17 minutes
  The measuring method of the pain is Electric pulp tester

SECONDARY OUTCOMES:
change from baseline in intensity of the pain | Change from Baseline up to 60 minutes
  using visual analog scale(VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Islamic Azad University, Tehran, Tehran Province, Iran